CLINICAL TRIAL: NCT02432053
Title: An Open Label, Multi-centre, Prospective Study to Demonstrate Safety and Efficacy of Once Daily Advagraf in Patients Undergoing Kidney or Liver Transplantation in India
Brief Title: A Study to Demonstrate Safety and Efficacy of Advagraf in Patients Undergoing Kidney or Liver Transplantation in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-0894; AS/111/10 (Other: Astellas Pharma India)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Transplantation; Liver Transplantation
Keywords: FK506; Advagraf; Tacrolimus; Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplantation (Experimental): Advagraf
  Interventions: Drug: Advagraf

INTERVENTIONS:
Drug: Advagraf
  Other Names: Modified release tacrolimus; FK506

SUMMARY:
The objective of the study is to demonstrate safety and efficacy of once-daily Advagraf in adult population undergoing kidney or liver transplantation in India.

DETAILED DESCRIPTION:
This is a phase IV, multi-centre, open label prospective study of once daily Advagraf in 200 patients undergoing kidney or liver transplantation in India. Adult patients undergoing kidney or liver transplantation and meeting all other eligibility criteria will be enrolled in the study. Enrolled patients will be administered once daily dose of Advagraf for 12 weeks. During these 12 weeks a total of 9 regular visits will be undertaken.

ELIGIBILITY:
Inclusion Criteria (common to kidney and liver transplant patients):

* Male or female patients between 18 to 65 years of age, undergoing liver or kidney transplantation
* Female patients of child bearing potential must have a negative serum pregnancy test prior to enrolment and must agree to practice effective birth control during the study. Tacrolimus may reduce the clearance of steroid based contraceptives leading to increased hormone exposure; particular care should be exercised when deciding upon contraceptive measures.
* Patients should be capable of understanding the purpose and risks of the study, and should provide written informed consent to participate in the study.

Inclusion Criteria (specifically for kidney transplant patients):

* Patients with end stage kidney disease and who are a suitable candidate for primary kidney transplantation.
* Patients scheduled to receive a kidney transplant from a cadaveric or living donor between 5 and 65 years of age with compatible ABO blood type.

Inclusion Criteria (specifically for liver transplant patients):

* Patients with end stage liver disease and who are a suitable candidate for primary liver transplantation.
* Patients scheduled to receive a liver transplant from a cadaveric or living donor between 5 and 65 years of age with compatible ABO blood type.

Exclusion Criteria (common to kidney and liver transplant patients):

* Previously received or are scheduled to receive an organ transplant other than kidney or liver
* Undergoing re-transplant from either a cadaveric or living donor
* Contraindication to the use of tacrolimus or corticosteroids.
* Malignancy or history of malignancy within the last 5 years, except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Systemic infection requiring treatment.
* Transplantation of kidney or liver from non-heart beating donor.
* Severe diarrhea, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus.
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the patient.
* Simultaneously participating in another investigational drug study or has participated in such study within 28 days prior to entry in this study.
* Receiving any non-registered medication or has received any non-registered medication within 28 days prior to entry in this study.
* Pregnant women or breast-feeding mother.
* Patients or respective donors known to be positive for human immunodeficiency virus (HIV).
* Unlikely to comply with the visits scheduled in the protocol.

Exclusion criteria (Specifically for kidney transplant patients)

* Cold ischemia time of the donor kidney > 30 hours.
* High immunological risk, defined as a positive cross match or PRA grade 50% in the previous 6 months.
* Liver cirrhosis.
* Significant liver disease, defined as having either elevated serum glutamic pyruvic transaminase / alanine aminotransferase(SGPT / ALT) (at least 2.5 times the upper value of the normal range at the investigational site) or elevated serum glutamic oxaloacetic transaminase/ aspartate transaminase (SGOT/AST) (at least 2.5 times the upper value of the normal range at the investigational site) or elevated total bilirubin levels (at least 2.5 times the upper value of the normal range at the investigational site) or all of them during the 28 days prior to entry into the study.
* Patients or respective donors known to be positive for hepatitis B virus (HBV) or hepatitis C virus (HCV).

Exclusion Criteria (specifically for liver transplant patients):

* Transplanted for hepatocellular carcinoma with a single nodule greater than 5.0 cm in diameter or more than 3 nodules or metastases or vascular tumoral invasion.
* Serum creatinine 2mg/dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Renal function (evaluated by level of Serum Creatinine) | from Day 0 to Week 12
Lipid profile | 0, 4, and 12-week
Incidence of New-Onset Diabetes Mellitus After Transplant (NODAT) | from Day 0 to Week 12
  NODAT is defined as a composite endpoint consisting of first occurrence of one of 4 parameters: (1) Two fasting plasma glucose (FPG) levels > 126 mg/dL which are > 30 days apart. (2) Oral hypoglycemic agent use for > 30 consecutive days. (3) Insulin therapy for > 30 consecutive days and (4) HbA1c > 6.5%
Incidence of infection | from Day 0 to Week 12
For kidney transplant patients: Event rate of patients with biopsy-confirmed acute rejections (BCAR) ≥ Grade I according to -The Banff 2007 working classification of renal allograft pathology within the first 12 weeks following kidney transplantation | from Day 0 to Week 12
  The biopsy shall be performed prior to the initiation of any anti-rejection therapy and as soon as possible after the onset of clinical / laboratory signs indicative of possible rejection
For liver transplant patients: Event rate of patients with biopsy-confirmed acute rejections (BCAR) with Rejection Activity Index of ≥ 4, within the first 12 weeks following liver transplantation | from Day 0 to Week 12
  The biopsy shall be performed prior to the initiation of any anti-rejection therapy and as soon as possible after the onset of clinical / laboratory signs indicative of possible rejection. Biopsy-confirmed acute rejections (BCAR) with Rejection Activity Index was defined according to The 1997 Banff schema for grading liver allograft rejection

SECONDARY OUTCOMES:
Time to first biopsy confirmed acute rejection episode | from Day 0 to Week 12
Overall frequency of acute rejection episodes | from Day 0 to Week 12
Severity of biopsy confirmed acute rejections | from Day 0 to Week 12
Incidence of corticosteroid resistant rejection | from Day 0 to Week 12
Incidence of corticosteroid sensitive rejection | from Day 0 to Week 12
Incidence of use of anti-lymphocyte antibodies | from Day 0 to Week 12
Graft loss | Week 12
Death | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- India (7):
  - Andhra Pradesh
  - Bangalore
  - Chennai
  - Mumbai
  - New Delhi
  - Tamil Nadu
  - Uttar Pradesh